CLINICAL TRIAL: NCT03439098
Title: Effects of Fermented Codonopsis Lanceolata on Improvement in Cognitive-Bio-Markers of Cognitive Functions in Healthy Adults With Subjective Memory Impairment: An 8-week Prospective Randomized Double-Blind Placebo-Controlled Trial With Multimodal Neuroimaging and Neurocognitive Assessments
Brief Title: Effects of Fermented Codonopsis Lanceolata on Improvement in Cognitive-Bio-Markers of Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EBI_CT_FCL
Record Dates: First submitted 2015-12-28; First posted 2018-02-20 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Subjective Memory Complaints

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fermented Codonopsis lanceolata 525mg (Experimental): Fermented Codonopsis lanceolata 525mg/day
  Interventions: Dietary Supplement: Fermented Codonopsis lanceolata 525mg
- Fermented Codonopsis lanceolata 1050mg (Experimental): Fermented Codonopsis lanceolata 1050mg/day
  Interventions: Dietary Supplement: Fermented Codonopsis lanceolata 1050mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented Codonopsis lanceolata 525mg — Fermented Codonopsis lanceolata 525mg daily for 8 weeks
  Arms: Fermented Codonopsis lanceolata 525mg
Dietary Supplement: Fermented Codonopsis lanceolata 1050mg — Fermented Codonopsis lanceolata 1050mg daily for 8 weeks
  Arms: Fermented Codonopsis lanceolata 1050mg
Dietary Supplement: Placebo — Placebo daily for 8 weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate the cognitive enhancement effect and safety of Fermented Codonopsis lanceolata, using the cognitive and clinical indicators (e.g. memory, attention, and psychomotor speed) and the latest brain imaging methods for healthy adults suffering subjective cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 65 years old
* Global Deterioration Scale score (GDS) of 2
* High school or higher levels of education
* With informed consent

Exclusion Criteria:

* Evidence of neurologic or medical conditions
* Axis I diagnosis when assessed by the board certified psychiatrist using the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorder, 4th edition (DSM-IV)(SCID-IV)
* Mini-mental status examination score of 25 or less
* Clinical Dementia Rating score of 0.5 or more suggesting cognitive impairment beyond self-perceived subjective deficits
* Intelligence quotient less than 70
* Any history of head trauma involving loss of consciousness or seizure
* Contraindications to magnetic resonance imaging (MRI)
* Use of psychotropics in last 3 months
* Allergic adverse reactions to Fermented Codonopsis lanceolata
* Participation in other clinical trials during the study period that might affect the outcome of the present study
* Use of oral contraceptive medication
* Current pregnancy or breast-feeding

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Changes in standardized scores on a neuropsychological test battery | baseline, 4th week, 8th week
  A composite z-scores were calculated from the scores of the neuropsychological test battery on attention and working memory. The test battery included Letter-number sequencing, Digit span (forward), and tasks from the Cambridge Neuropsychological Test Automated Battery (CANTAB) including the Match-to-Sample Visual Search, Reaction Rime, Rapid Visual Information Processing, and Stop Signal tasks.

SECONDARY OUTCOMES:
Changes in scores of the Subjective Memory Complaints Questionnaire | baseline, 4th week, 8th week
  The Subjective Memory Complaints Questionnaire (SMCQ) contains 14 items and consists of two domains: global memory function and everyday memory function. The response to each item is rated as "yes" (1 point) or "no" (0 point). The total score ranges from 0 to 14 points, and higher points indicate larger degrees of subjective memory complaints.
Number of participants with adverse events | 4th week, 8th week
Changes of brain volume in magnetic resonance imaging assessed by computational approaches | baseline, 8th week
  Volumes of the clusters in the brain are reported in cubic millimeters
Changes of cortical thickness in magnetic resonance imaging assessed by computational approaches | baseline, 8th week
  Cortical thickness is measured in millimeters.
Functional brain changes in magnetic resonance imaging assessed by computational approaches | baseline, 8th week
  The Blood Oxygenation Level Dependent (BOLD) signal intensities in arbitrary units are measured in each voxel of the brain. These values are compared between the time points and groups, and the statistical values are presented as results.
Metabolic brain changes in magnetic resonance imaging assessed by computational approaches | baseline, 8th week
  Brain metabolite concentrations are assessed using the magnetic resonance spectroscopy and are estimated in mmol per liter.

CONTACTS AND LOCATIONS:
Overall Officials: Inkyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ewha Womans University
Locations (1):
- Ewha Womans University, Seoul, South Korea